CLINICAL TRIAL: NCT03822312
Title: A Pilot Study of Digital Breast Tomosynthesis Guided Near-infrared Tomographic Optical Breast Imaging (DBT-TOBI) in Monitoring Response of Breast Cancer to Neoadjuvant Therapy
Brief Title: A Pilot Study of Tomographic Optical Breast Imaging (DBT-TOBI) to Monitor Response to Neoadjuvant Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven J Isakoff, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-333; 1R01CA187595 (NIH)
Record Dates: First submitted 2018-12-22; First posted 2019-01-30 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Optical imaging; neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- DBT-TOBI (Experimental): * Subjects will be imaged using DBT-TOBI at the time points indicated in the Study Calendar (Baseline, before cycle 2, and additional optional time points).
  * Both breasts will be measured in turn.
  * Each breast is symmetrically centered on the x-ray detector/optical illuminator and is first compressed according to standard mammography procedures to determine the amount of force needed for each given patient
  * An optional Magnetic Resonance Imaging TOBI (MRI-TOBI) scan will also be performed.
  Interventions: Device: DBT-TOBI; Device: MRI-TOBI

INTERVENTIONS:
Device: DBT-TOBI — The DBT-TOBI scan system is designed to deliver low power laser lights through a person's body tissue and collect data about the light that is transmitted through
Device: MRI-TOBI — The MRI-TOBI scan system is designed to deliver low power laser lights through a person's body tissue and collect data about the light that is transmitted through. The MRI scan is completed at the same time as the TOBI scan. Participation in this part of the intervention is optional.

SUMMARY:
This research study is evaluating whether the use of digital breast tomosynthesis and near-infrared tomographic optical breast imaging (DBT-TOBI) scans can predict the response of triple negative or HER2+ breast cancer to neoadjuvant chemotherapy.

The study radiologic scan involved in this study is digital breast tomosynthesis (also called 3 Dimensional mammogram) combined with near-infrared tomographic optical breast imaging, or DBT-TOBI.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study device for this indication.

The FDA (the U.S. Food and Drug Administration) has not approved DBT-TOBI as a diagnostic scan for this disease.

The DBT-TOBI scan system is designed to deliver low power laser lights through a person's body tissue and collect data about the light that is transmitted through. In this study, the DBT-TOBI will be used to scan the breast. The data that can be collected through the scan is the total hemoglobin concentration and hemoglobin oxygen saturation. Hemoglobin is the protein found in red blood cells that is responsible for carrying oxygen to the various tissues in the body. These two data types are thought to provide insight into the response of the breast cancer to neoadjuvant chemotherapy treatment response. The researchers are looking to find if these scans will help show changes in the hemoglobin levels, thus showing how the cancer is reacting to treatment. The study is focused on 2 types of breast cancer called triple negative breast cancer and Human Epidermal Growth Factor Receptor 2 (HER2).

ELIGIBILITY:
Inclusion Criteria:

* Female
* Participant will be receiving neoadjuvant chemotherapy at the Massachusetts General Hospital (MGH) Center for Breast Cancer.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured as ≥10 mm in the longest diameter with breast MRI, mammography or ultrasound. See Section 11 for the evaluation of measurable disease.
* Patients must have Humane Epidermal Growth Factor Receptor (HER2) positive (regardless of Hormone Receptor (HR) status) or Triple Negative (TN) disease as confirmed by pathology. HER2 positive is defined according to ASCO-CAP guidelines, and patient will be receiving HER2 directed therapy. TN is defined as Estrogen Receptor <=1%, Progesterone Receptor <= 1%, and HER2 negative by American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines. For tumors with discordant or borderline receptor findings, the Principal Investigator will adjudicate the final decision.
* Age 18 and above.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with open wounds on the breast.
* Patients who have undergone breast surgery or breast biopsy 10 days or less prior to the first planned optical imaging scan.
* Patients with breast implants.
* Patients whose primary lesion is outside the field of view of the optical imaging system.
* A history of ipsilateral disease (including invasive breast cancer, ductal carcinoma in situ (DCIS), and benign lesions) or breast surgery.
* Patients who are pregnant or trying to become pregnant.
* Medical or psychiatric conditions which, in the opinion of the investigator, might result in risk to the subject from participation in the study or inability to complete the study.
* For patients who agree to participate in the optional MRI study, these following additional exclusion criteria also apply:

  * Neurostimulators;
  * Pacemakers;
  * Implanted metallic material or devices (metal implants or large tattoos in the field of view);
  * Severe claustrophobia;
  * Physical characteristics (weight and/or size) that exceed the capabilities of the MRI scanner;
  * Known allergy or hypersensitivity reactions to gadolinium, versetamide, or any of the inert ingredients in gadolinium-based contrast agents;
  * Severe renal insufficiency, e.g., estimated glomerular filtration rate < 30 mL/min.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determining whether DBT-TOBI total hemoglobin concentration measurements before cycle 3 of chemotherapy can predict pathological complete response (pCR) versus non-complete responses in breast cancer. | 4 to 6 months
  The primary aim is to evaluate whether early measurements of the total hemoglobin concentration ratio in the primary tumor vs. the surrounding tissue, as estimated by our DBT-TOBI system, can predict neoadjuvant chemotherapy response at the time of surgery. Measurements will be obtained at baseline and just before cycle 3 to determine whether DBT-TOBI is predictive of pathological complete response (pCR) versus non-complete response for Human Epidermal Growth Factor Receptor 2 (HER2) positive and Triple negative breast cancer patients undergoing neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Determining the predictive performance of early DBT-TOBI scans before the 3rd cycle of chemotherapy in distinguishing pCR versus non-pCR based on changes in tissue hemoglobin oxygen saturation. | 4-6 months
  DBT-TOBI measurements of the changes in the ratio of hemoglobin oxygen saturation in the primary tumor versus surrounding normal area between the pre-treatment baseline and immediately before the 3rd cycle of therapy will be used to predict pathological outcome at surgery. The outcome will be quantified using the area under the curve (AUC) after estimating an empirical receiver operating characteristic (ROC) curve for predicting pCR vs non-pCR.
Determining whether other optical parameters measured by DBT-TOBI are predictive of the final pathologic response after neoadjuvant therapy. | 4-6 months
  DBT-TOBI will be used to measure changes in the ratio of tumor to normal hemoglobin oxygen saturation ratio (SO2,T/N) between the baseline and prior to cycle 3 scans, as well as changes in the temporal response of total hemoglobin concentration (HbTT/N) or oxygen saturation (SO2,T/N) under constant mammographic compression.
Determining whether DBT-TOBI total hemoglobin concentration measurements before the cycle 2 and after changing chemotherapy can predict pathological complete response (pCR) versus non-complete responses in breast cancer. | 4-6 months
  DBT-TOBI measurements of the changes in the ratio of total hemoglobin concentration in the primary tumor versus surrounding normal area between the pre-treatment baseline and immediately before the 2nd cycle of therapy and immediately before any change in chemotherapy will be used to predict pathological outcome at surgery.
To investigate the ability of DBT-TOBI measurements to predict Residual Cancer Burden (RCB) groups 0 and 1 versus 2 and 3. | 4-6 months
  The various DBT-TOBI measurements (including the changes in the ratio of total hemoglobin concentration or oxygen saturation in the primary tumor versus surrounding normal area) between the pre-treatment baseline and immediately before the 3rd cycle of therapy and immediately before any change in chemotherapy will be used to predict pathological outcome at surgery. For this objective, the Residual Cancer Burden (RCB) categorization will be used and RCB 0/1 will be compared to RCB 2/3.
To investigate whether compression response-based optical property metrics are associated with lesion stiffness as measured by Magnetic Resonance Elastography. | 4-6 months
  The DBT-TOBI measurements under mammographic compression will be used to compare to the the measurements of tumor stiffness by Magnetic Resonance Imaging elastography. These measurements will be made at baseline and before the 3rd cycle of chemotherapy.
To assess the threshold values for detecting pathologic Complete Response (pCR) versus non-PCR and Residual Cancer Burden (RCB) 0/1 versus RCB 2/3, respectively, for changes in optical parameters at standard time points. | 4-6 months
  For this aim, a Receiver Operator Curve (ROC) will be estimated and used to determine the optimum cut-off value of optical parameters measured by DBT-TOBI from baseline to just prior to the 2nd or 3rd therapy cycle of chemotherapy, and from just before any chemotherapy change to just before the 2nd cycle with the second agent (as applicable), that distinguishes pCR from non-pCR and separately for RCB 0/1 from RCB 2/3.
To assess the threshold values for detecting pCR vs. non-PCR and RCB 0/1 versus RCB 2/3, respectively, for changes in MR derived tumor morphology from baseline to just prior the 3rd therapy cycle. | 4-6 months
  For this aim, a Receiver Operator Curve (ROC) will be estimated and used to determine the optimum cut-off value of MR derived tumor morphology from baseline to just prior to the 2nd or 3rd therapy cycle of chemotherapy, and from just before any chemotherapy change to just before the 2nd cycle with the second agent (as applicable), that distinguishes pCR from non-pCR and separately for RCB 0/1 from RCB 2/3.
To compare the predictive abilities between the Receiver Operator Curve (ROC) developed using DBT-TOBI and MR derived tumor morphology measurements to determine which measure more accurately predicts pathologic response. | 4-6 months
  For this aim, the Receiver Operator Curves (ROC) developed in Outcome 7 (using DBT-TOBI optical parameters) and 8 (using MR derived tumor morphology) will be compared and the difference will be used to determine which measure more accurately identifies patients with pCR vs non-PCR and patients with RCB 0/1 versus RCB 2/3.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Isakoff, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor- Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Requests may be directed to: [contact information for Sponsor- Investigator or designee].